CLINICAL TRIAL: NCT06334757
Title: A Multi-center, Open-label, Single-arm Study to Evaluate the Efficacy and Safety of Serplulimab Plus Bevacizumab and Chemotherapy for EGFRm+ Locally Advanced or Metastasis Non-Squamous NSCLC Patients After EGFR-TKI Treatment Failure
Brief Title: Serplulimab Plus Bevacizumab and Chemotherapy for EGFR-mutant Metastatic NSCLC Patients After EGFR-TKI Treatment Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX10IIT22
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2023-04

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serplulimab+Bevacizumab+Pemetrexed+Carboplatin (Experimental): Using Serplulimab in combination with bevacizumab, carboplatin and pemetrexed to treat patients with EGFR mutated, advanced non-small cell lung cancer (NSCLC) after failure of EGFR tyrosine kinase inhibitors.
  Interventions: Drug: Serplulimab; Drug: Bevacizumab Biosimilar HLX04; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Serplulimab — 300 mg，IV，Q3W
  Other Names: HLX10
Drug: Bevacizumab Biosimilar HLX04 — 7.5 mg/kg，Q3W
  Other Names: HLX04
Drug: Pemetrexed — 500 mg/m2，IV，Q3W
Drug: Carboplatin — AUC=5，IV，Q3W

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Serplulimab Plus Bevacizumab and chemotherapy in TKI-resistant EGFR-mutated non-squamous NSCLC Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent before any trial-related processes;
2. Age ≥ 18 years and ≤70 years male or females;
3. Has a histologically or cytologically confirmed stage IIIB/IIIC (American Joint Committee on Cancer [AJCC] 8th edition) NSCLC that is unresectable and not fit for radical concurrent chemoradiotherapy, or metastatic / recurrent non-squamous NSCLC;
4. Patients with EGFR mutation confirmed by tumor histology or cytology or hematology prior to EGFR-TKI treatment
5. EGFR-TKI resistance, confirmed by RECIST 1.1
6. The Eastern Cancer Cooperative Group (ECOG) performance score of 0 or 1;

Exclusion Criteria:

1. History of severe allergies to any study drug
2. Has previously received the following therapies: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or any other stimulatory or inhibitory agents of T cell receptors
3. Previous exposure to VEGF inhibitor for anti-cancer treatment
4. Patients with untreated symptomatic brain metastases. Patients with treated brain metastases will be allowed if brain imaging obtained greater than 4 weeks from trial enrollment reveals stable disease.
5. Has received a live-virus vaccination within 28 days of planned treatment start
6. Interstitial lung disease or pneumonitis requiring oral or IV glucocorticoids Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR(Overall Response Rate) | From start of treatment to 12 months
  The proportion of subjects who have a complete response (CR) or a partial response (PR)

SECONDARY OUTCOMES:
PFS(Progression Free Survival) | From start of treatment to 24 months
  Time from enrollment to first disease progression assessed by investigator or death due to any cause
OS(Overall Survival) | From start of treatment to 24 months
  Time from enrollment to the death of the subject due to any cause
AE(Adverse Event) | From start of treatment to 24 months
  incidece of adverse drug event

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China